CLINICAL TRIAL: NCT01924143
Title: An Open-Label Study to Evaluate the Absorption, Distribution, Metabolism, and Excretion of TD-9855 Following a Single Oral Dose Containing Approximately 100 µCi [14C]-Labeled TD-9855 (20 mg) in Healthy Subjects
Brief Title: TD-9855 Mass Balance Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0105
Record Dates: First submitted 2013-08-09; First posted 2013-08-16 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: ADHD; Fibromyalgia
Keywords: ADHD; Fibromyalgia
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Fibromyalgia | interventions — ampreloxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TD-9855 (Experimental)
  Interventions: Drug: TD-9855

INTERVENTIONS:
Drug: TD-9855 — radiolabeled (100 µCi [14C]-Labeled) TD-9855 (20 mg)

SUMMARY:
The purpose of the study is to evaluate the absorption, distribution, metabolism, and excretion (ADME) of a single oral dose of [14C]TD-9855

ELIGIBILITY:
Inclusion Criteria:

* Healthy, nonsmoking male subjects or healthy, nonsmoking female subjects not of childbearing potential, 18 to 50 years old, inclusive. Women are considered to be not of childbearing potential if they have had a hysterectomy or tubal ligation or are at least 2 years postmenopausal (follicle-stimulating hormone [FSH] >40 IU/mL)
* Body mass index 19 to 31 kg/m2, inclusive, and weight at least 55 kg
* Negative for hepatitis B, hepatitis C, and HIV antibody

Exclusion Criteria:

* Have evidence or history of clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of dosing), hematological, endocrine, dermatologic, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease
* Subjects who, in the opinion of the investigator, are at risk for suicide or risk of harming others, or who score positive on the C-SSRS (item 2 or higher on ideation). Subjects with any history of suicide attempts
* Any condition possibly affecting drug absorption (e.g., previous surgery on the gastrointestinal tract [including removal of parts of the stomach, bowel, liver, gall bladder, or pancreas])
* Infrequent bowel movements (less than once per 24 hours) in the last 7 days prior to Day -1. Subject is unable to provide a fecal sample prior to study drug dosing on Day -1 or Day 1.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To define the routes and rates of elimination and mass balance of [14C]-labeled TD-9855 | 1-21 Days
  Urinary and fecal recovery of total radioactivity. Whole blood and plasma concentrations of total radioactivity.

SECONDARY OUTCOMES:
Pharmacokinetics of total drug-related material and TD-9855: Cmax | 1-21 Days
  Whole blood and plasma concentrations
PK: Tmax | 1-21 Days
  Whole blood and plasma concentrations
PK: AUCt | 1-21 Days
  Whole blood and plasma concentrations
PK: AUCinf | 1-21 Days
PK: CL/F (Renal clearance) | 1-21 Days
  Urine
PK: Vz/F (oral volume of distribution during the terminal phase) | 1-21 Days
PK: amount excreted in urine (Ae) | 1-21 Days
  Urine
PK: CLR (Renal clearance, computed as amount recovered in urine/ AUCinf) | 8-21 Days
  Urine
Metabolic profiles in plasma and excreta | 1-21 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.